CLINICAL TRIAL: NCT03838016
Title: Babble Boot Camp: Preventing Speech and Language Disorders in Children With Classic Galactosemia
Brief Title: Preventing Speech and Language Disorders in Children With Classic Galactosemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Washington State University (Other)
Responsible Party: Principal Investigator, Beate Peter, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004969
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2024-09

CONDITIONS: Classic Galactosemia; Speech Disorders in Children; Language Disorders in Children
MeSH Terms: conditions — Galactosemias

STUDY DESIGN:
Intervention Model Description: The investigators created an intervention program, Babble Boot Camp (BBC), designed to support communication skills during the prespeech and early speech and language stages. One cohort with classic galactosemia (CG) enters this treatment at age 2-5 months and is monitored closely using audio and video recordings and questionnaires. A second cohort with CG enters close monitoring at age 2-5 months but starts treatment at age 15 months. A typical cohort enters close monitoring at age 2-5 months. Treatment and close monitoring ends at age 24 months. Follow-up testing of speech and language skills and questionnaire data about child development and parent well-being is collected once a year at ages 2 ½, 3 ½, and 4 ½ years. A cohort with CG, age 6 months to 4 ½ years, too old for any treatment and close monitoring, provides the same data as the other cohorts at ages 2 ½, 3 ½, and 4 ½ years. Results will show whether the BBC is effective and, if yes, which start age is best.
Who Masked: Outcomes Assessor
Masking Description: Team members who conduct assessments or analyze data do not have access to a child's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment cohort with classic galactosemia (Experimental): These children and their parents receive the Babble Boot Camp intervention and also participate in the close monitoring activities (progress reports that the speech-language pathologist generates during the online meeting with the family; monthly daylong audio recording; questionnaires that are sent out every three to six months; formal speech and language testing at ages 2 1/2, 3 1/2, and 4 1/2 years).
  Interventions: Behavioral: Babble Boot Camp
- Treatment cohort with classic galactosemia, delayed start (Experimental): The children in the control cohort enter the study when they are younger than 5 months old and participate in the close monitoring until they are 24 months old. They start getting the same treatment type and intensity as the treatment cohort but at a delayed age, when they turn 15 months.
  Interventions: Behavioral: Babble Boot Camp
- Older control cohort with classic galactosemia (No Intervention): The children in the older control cohort are 6 months to 4 1/2 years old and provide standardized test results in the area of speech and language development at child ages 2 1/2, 3 1/2, and 4 1/2 years. They receive no treatment and no close monitoring. These families provide questionnaire information every three months until child age 24 months.
- Typical controls (No Intervention): These children are free of any medical or developmental diagnosis. They enter the study at ages 2 to 5 months and provide close monitoring data until they are 24 months old, then they receive standardized speech and language testing at ages 2 1/2, 3 1/2, and 4 1/2 years, just like the treatment cohort, but the typical controls receive no treatment under this study.

INTERVENTIONS:
Behavioral: Babble Boot Camp — The Babble Boot Camp is an experimental study to investigate whether earliest and proactive activities and routines can positively influence the speech and language development of children who were diagnosed with classic galactosemia at birth. A speech-language pathologists implements the intervention by teaching parents to foster and expand earliest signals of communication, prespeech activities such as coo and babble, vocabulary growth, sentence complexity, and use of language to communicate. Examples are intentional eye contact, reinforcing babble with rewarding play activities, and repeating a child's rudimentary sentence with slight expansions to scaffold longer sentences.
  Arms: Treatment cohort with classic galactosemia; Treatment cohort with classic galactosemia, delayed start

SUMMARY:
A critical knowledge gap is whether proactive intervention can improve speech and language outcomes in infants at known risk for communication disorders. Speech and language assessments and treatments are usually not initiated until deficits can be diagnosed, no earlier than age 2-3 years. Preventive services are not available. Children with classic galactosemia (CG) hold the keys towards investigating whether proactive services are more effective than conventional management. CG is a recessively inherited inborn error of metabolism characterized by defective conversion of galactose. Despite early detection and strict adherence to lactose-restricted diets, children with CG are at very high risk not only for motor and learning disabilities but also for severe speech sound disorder and language impairment. Delays are evident from earliest signals of communication and persist into adulthood in many cases but speech/language assessment and treatment are usually not initiated until deficits manifest. However, because CG is diagnosed via newborn screening, the known genotype-phenotype association can be leveraged to investigate the efficacy of proactive interventions during the acquisition of prespeech (2 to 12 months) and early communication skills (13 to 24 months). If this proactive intervention is more effective than standard care regarding speech and language outcomes in children with CG, this will change their clinical management from deficit-based to proactive services. It will also motivate investigating this approach in infants with other types of known risk factors, e.g., various genetic causes and very low birth weight.

The Babble Boot Camp is a program for children with CG, ages 2 to 24 months. The intervention is implemented by a pediatric speech-language pathologist (SLP) via parent training. Activities and routines are designed to foster earliest signals of communication, increase coo and babble behaviors, support the emergence of first words and word combinations, and expand syntactic complexity. The SLP meets with parents online every week for 10 to 15 minutes to provide instruction, feedback, and guidance. Close monitoring of progress is achieved via regularly administered questionnaires, a monthly day-long audio recording, and the SLPs weekly progress notes. At age 24 months, the active phase of the Babble Boot Camp ends. The children receive a professional speech/language assessment at ages 2 1/2, 3 1/2, and 4 1/2 years.

DETAILED DESCRIPTION:
Speech and language assessments and treatments are usually not initiated until deficits can be diagnosed, which occurs at age 2-3 years at the earliest. Preventive services are not available. Children with classic galactosemia (CG) hold the keys towards investigating whether proactive services are more effective than conventional management. CG is a recessively inherited inborn error of metabolism characterized by defective conversion of galactose. Despite early detection and strict adherence to lactose-restricted diets, children with CG are at very high risk not only for motor and learning disabilities but also for severe speech sound disorder and language impairment. Delays are evident from earliest signals of communication and persist into adulthood in many cases. As with most other children, speech and language assessments and treatment are usually not initiated until deficits manifest. However, because CG is diagnosed via newborn screening, the known genotype-phenotype association can be leveraged to investigate whether proactive interventions during the acquisition of prespeech (2 to 12 months) and early communication skills (13 to 24 months) can mitigate the speech and language deficits. If the investigators show that interventions during the first two years of life are more effecting in improving speech and language outcomes in children with CG, compared to traditional care, this will change their clinical management from deficit-based to proactive services. It will also motivate investigating this approach in infants with other types of known risk factors for communication disorders, e.g., various genetic causes and very low birth weight.

The investigators created an intervention program designed to support communication abilities during the prespeech and early speech and language stages for ages 2 to 24 months. The Babble Boot Camp (BBC) is implemented via parent training by a speech-language pathologist (SLP) with expertise in early childhood using Zoom, a HIPAA-compliant telepractice software provided for free by the PI's institution, to connect with the families. Zoom runs on computers, tablets, and smartphones. Parents learn about the typical milestones of prespeech, speech, and language development, potential red flags for delays, and importantly, activities that support typical development for all stages of the program. Following an orientation to the program, the SLP meets with each family once per week for training and consultation the relevant activities given the child's current speech/language status. Examples of activities are stimulating and reinforcing coos and babble, enriching the child's linguistic environment with joint book reading and pointing out the names of objects, and expanding child utterances to provide slightly more complex model sentences. The key principle underlying all activities is the zone of proximal development, also referred to as scaffolding, where parents provide speech and language models that bridge what the child can already to and what is slightly beyond the child's skill set: the model is in the zone of skills that the child can do with help. One key skill that is targeted throughout the program is imitation. The program brochure includes the rationale, instructions, and examples for each activity, such as (direct quote from the brochure): "Expanding on your child's utterance will provide a model for more complex sentence structures as well as increase her/his vocabulary. An added benefit is to let your child hear words in their correctly produced forms when her/his own productions are showing some incorrect speech sounds. This will build your child's awareness of what the word should sound like and get her/him ready to try the correct form. Throughout your daily routine, listen to your child's utterances and expand upon them slightly. You can add descriptive words or fill in some missing words to make a more complete sentence without overwhelming your child's ability to comprehend your sentence.

Examples: Child: "Goggie bye-bye." Parent: "Yeah, that doggie is going bye-bye!" - Child:

"Mommy doing?" Parent: "What is Mommy doing? She is taking Sammie outside."

ELIGIBILITY:
Inclusion Criteria:

* Newborn diagnosis of classic galactosemia
* Any ethnic or racial background
* Primary language in the home is English
* Any geographic region in the US and other countries because the intervention is done online
* Computer and internet access (we can help if a family wants to participate but doesn't have this access)
* At least one parent must have at least an 8th grade education to be able to fill out the questionnaires

Exclusion Criteria:

* Other forms of galactosemia outside of classic galactosemia
* Medical, sensory, or psychiatric condition that could introduce confounding, e.g., Trisomy 21 or deafness

Ages: 2 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 285 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Speech sound production accuracy | Through study completion, an average of 4 years 2 months
  Standardized testing of speech sounds using a published test of articulation
Expressive language skills | Through study completion, an average of 4 years 2 months
  Standardized testing of expressive language ability, using a published test of child language

SECONDARY OUTCOMES:
Cognitive development | Through study completion, an average of 4 years 2 months
  Standardized testing of cognitive development, using a published test
Quality of life using the PedsQL questionnaires | Through study completion, an average of 4 years 2 months
  Questionnaire-based assessment of quality of life for the child and parent(s). Captures physical functioning, physical symptoms, emotional functioning, social functioning, and cognitive functioning for children. Captures physical functioning, emotional functioning, social functioning, and work/school function for adults.
Child health and development using the Ages and Stages Questionnaires 3 | Through study completion, an average of 4 years 2 months
  Questionnaire-based assessment of child development in the areas of communication, gross motor, fine motor, problem solving, and personal-social development for children.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified. Only data that are reported in publications will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared at the time of publication of results, no end date.
Access Criteria: Qualified researchers will be given access to the de-identified data. These are researchers who provide a methodologically sound proposal

REFERENCES:
- [Background] Demirbas D, Coelho AI, Rubio-Gozalbo ME, Berry GT. Hereditary galactosemia. Metabolism. 2018 Jun;83:188-196. doi: 10.1016/j.metabol.2018.01.025. Epub 2018 Jan 31. PMID 29409891
- [Background] Antshel KM, Epstein IO, Waisbren SE. Cognitive strengths and weaknesses in children and adolescents homozygous for the galactosemia Q188R mutation: a descriptive study. Neuropsychology. 2004 Oct;18(4):658-64. doi: 10.1037/0894-4105.18.4.658. PMID 15506833
- [Background] Potter NL, Nievergelt Y, Shriberg LD. Motor and speech disorders in classic galactosemia. JIMD Rep. 2013;11:31-41. doi: 10.1007/8904_2013_219. Epub 2013 Apr 2. PMID 23546812
- [Background] Waisbren SE, Norman TR, Schnell RR, Levy HL. Speech and language deficits in early-treated children with galactosemia. J Pediatr. 1983 Jan;102(1):75-7. doi: 10.1016/s0022-3476(83)80292-3. No abstract available. PMID 6848731
- [Background] Timmers I, van den Hurk J, Di Salle F, Rubio-Gozalbo ME, Jansma BM. Language production and working memory in classic galactosemia from a cognitive neuroscience perspective: future research directions. J Inherit Metab Dis. 2011 Apr;34(2):367-76. doi: 10.1007/s10545-010-9266-4. Epub 2011 Feb 3. PMID 21290187
- [Background] Lewis FM, Coman DJ, Syrmis M, Kilcoyne S, Murdoch BE. Charting a seven-year trajectory of language outcomes for a child with galactosemia. J Dev Behav Pediatr. 2013 Jul-Aug;34(6):414-8. doi: 10.1097/DBP.0b013e31829a7be1. PMID 23838587
- [Background] Lewis FM, Coman DJ, Syrmis M, Kilcoyne S, Murdoch BE. Differential phonological awareness skills in children with classic galactosemia: a descriptive study of four cases. JIMD Rep. 2013;10:45-52. doi: 10.1007/8904_2012_200. Epub 2012 Dec 29. PMID 23430800
- [Background] Potter NL, Lazarus JA, Johnson JM, Steiner RD, Shriberg LD. Correlates of language impairment in children with galactosaemia. J Inherit Metab Dis. 2008 Aug;31(4):524-32. doi: 10.1007/s10545-008-0877-y. Epub 2008 Jul 12. PMID 18649009
- [Background] Waggoner DD, Buist NR, Donnell GN. Long-term prognosis in galactosaemia: results of a survey of 350 cases. J Inherit Metab Dis. 1990;13(6):802-18. doi: 10.1007/BF01800204. PMID 1706789
- [Background] Storkel HL, Komesidou R, Fleming KK, Romine RS. Interactive Book Reading to Accelerate Word Learning by Kindergarten Children With Specific Language Impairment: Identifying Adequate Progress and Successful Learning Patterns. Lang Speech Hear Serv Sch. 2017 Apr 20;48(2):108-124. doi: 10.1044/2017_LSHSS-16-0058. PMID 28419188
- [Background] Dimitrova N, Ozcaliskan S, Adamson LB. Parents' Translations of Child Gesture Facilitate Word Learning in Children with Autism, Down Syndrome and Typical Development. J Autism Dev Disord. 2016 Jan;46(1):221-231. doi: 10.1007/s10803-015-2566-7. PMID 26362150
- [Background] Hassink JM, Leonard LB. Within-treatment factors as predictors of outcomes following conversational recasting. Am J Speech Lang Pathol. 2010 Aug;19(3):213-24. doi: 10.1044/1058-0360(2010/09-0083). Epub 2010 Mar 22. PMID 20308290
- [Background] Roy BC, Frank MC, DeCamp P, Miller M, Roy D. Predicting the birth of a spoken word. Proc Natl Acad Sci U S A. 2015 Oct 13;112(41):12663-8. doi: 10.1073/pnas.1419773112. Epub 2015 Sep 21. PMID 26392523
- [Background] Oller DK, Niyogi P, Gray S, Richards JA, Gilkerson J, Xu D, Yapanel U, Warren SF. Automated vocal analysis of naturalistic recordings from children with autism, language delay, and typical development. Proc Natl Acad Sci U S A. 2010 Jul 27;107(30):13354-9. doi: 10.1073/pnas.1003882107. Epub 2010 Jul 19. PMID 20643944
- [Background] Xu D, Richards JA, Gilkerson J. Automated analysis of child phonetic production using naturalistic recordings. J Speech Lang Hear Res. 2014 Oct;57(5):1638-50. doi: 10.1044/2014_JSLHR-S-13-0037. PMID 24824489
- [Background] Gilkerson J, Richards JA, Warren SF, Montgomery JK, Greenwood CR, Kimbrough Oller D, Hansen JHL, Paul TD. Mapping the Early Language Environment Using All-Day Recordings and Automated Analysis. Am J Speech Lang Pathol. 2017 May 17;26(2):248-265. doi: 10.1044/2016_AJSLP-15-0169. PMID 28418456
- [Background] Dykstra JR, Sabatos-Devito MG, Irvin DW, Boyd BA, Hume KA, Odom SL. Using the Language Environment Analysis (LENA) system in preschool classrooms with children with autism spectrum disorders. Autism. 2013 Sep;17(5):582-94. doi: 10.1177/1362361312446206. Epub 2012 Jul 2. PMID 22751753
- [Background] VanDam M, Oller DK, Ambrose SE, Gray S, Richards JA, Xu D, Gilkerson J, Silbert NH, Moeller MP. Automated Vocal Analysis of Children With Hearing Loss and Their Typical and Atypical Peers. Ear Hear. 2015 Jul-Aug;36(4):e146-52. doi: 10.1097/AUD.0000000000000138. PMID 25587667
- [Background] Caskey M, Stephens B, Tucker R, Vohr B. Importance of parent talk on the development of preterm infant vocalizations. Pediatrics. 2011 Nov;128(5):910-6. doi: 10.1542/peds.2011-0609. Epub 2011 Oct 17. PMID 22007020
- [Background] Soderstrom M, Wittebolle K. When do caregivers talk? The influences of activity and time of day on caregiver speech and child vocalizations in two childcare environments. PLoS One. 2013 Nov 18;8(11):e80646. doi: 10.1371/journal.pone.0080646. eCollection 2013. PMID 24260443
- [Background] Zimmerman FJ, Gilkerson J, Richards JA, Christakis DA, Xu D, Gray S, Yapanel U. Teaching by listening: the importance of adult-child conversations to language development. Pediatrics. 2009 Jul;124(1):342-9. doi: 10.1542/peds.2008-2267. PMID 19564318
- [Background] Welling L, Waisbren SE, Antshel KM, Colhoun HO, Gautschi M, Grunewald S, Holman R, van der Lee JH, Treacy EP, Bosch AM. Systematic Review and Meta-analysis of Intelligence Quotient in Early-Treated Individuals with Classical Galactosemia. JIMD Rep. 2017;37:115-123. doi: 10.1007/8904_2017_22. Epub 2017 Apr 9. PMID 28391442
- [Background] Schonhaut L, Armijo I, Schonstedt M, Alvarez J, Cordero M. Validity of the ages and stages questionnaires in term and preterm infants. Pediatrics. 2013 May;131(5):e1468-74. doi: 10.1542/peds.2012-3313. Epub 2013 Apr 29. PMID 23629619
- [Background] ten Hoedt AE, Maurice-Stam H, Boelen CC, Rubio-Gozalbo ME, van Spronsen FJ, Wijburg FA, Bosch AM, Grootenhuis MA. Parenting a child with phenylketonuria or galactosemia: implications for health-related quality of life. J Inherit Metab Dis. 2011 Apr;34(2):391-8. doi: 10.1007/s10545-010-9267-3. Epub 2011 Feb 3. PMID 21290186
- [Background] Robbins J, Klee T. Clinical assessment of oropharyngeal motor development in young children. J Speech Hear Disord. 1987 Aug;52(3):271-7. doi: 10.1044/jshd.5203.271. PMID 3455449
- [Result] Peter B, Potter N, Davis J, Donenfeld-Peled I, Finestack L, Stoel-Gammon C, Lien K, Bruce L, Vose C, Eng L, Yokoyama H, Olds D, VanDam M. Toward a paradigm shift from deficit-based to proactive speech and language treatment: Randomized pilot trial of the Babble Boot Camp in infants with classic galactosemia. F1000Res. 2019 Mar 11;8:271. doi: 10.12688/f1000research.18062.5. eCollection 2019. PMID 32566130
- [Result] Peter B, Davis J, Cotter S, Belter A, Williams E, Stumpf M, Bruce L, Eng L, Kim Y, Finestack L, Stoel-Gammon C, Williams D, Scherer N, VanDam M, Potter N. Toward Preventing Speech and Language Disorders of Known Genetic Origin: First Post-Intervention Results of Babble Boot Camp in Children With Classic Galactosemia. Am J Speech Lang Pathol. 2021 Nov 4;30(6):2616-2634. doi: 10.1044/2021_AJSLP-21-00098. Epub 2021 Oct 19. PMID 34665663
- [Result] Peter B, Davis J, Finestack L, Stoel-Gammon C, VanDam M, Bruce L, Kim Y, Eng L, Cotter S, Landis E, Beames S, Scherer N, Knerr I, Williams D, Schrock C, Potter N. Translating principles of precision medicine into speech-language pathology: Clinical trial of a proactive speech and language intervention for infants with classic galactosemia. HGG Adv. 2022 May 20;3(3):100119. doi: 10.1016/j.xhgg.2022.100119. eCollection 2022 Jul 14. PMID 35677809
- [Result] Finestack LH, Potter N, VanDam M, Davis J, Bruce L, Scherer N, Eng L, Peter B. Feasibility of a Proactive Parent-Implemented Communication Intervention Delivered via Telepractice for Children With Classic Galactosemia. Am J Speech Lang Pathol. 2022 Nov 16;31(6):2527-2538. doi: 10.1044/2022_AJSLP-22-00107. Epub 2022 Oct 14. PMID 36251874
- [Result] Peter B, Bruce L, Finestack L, Dinu V, Wilson M, Klein-Seetharaman J, Lewis CR, Braden BB, Tang YY, Scherer N, VanDam M, Potter N. Precision Medicine as a New Frontier in Speech-Language Pathology: How Applying Insights From Behavior Genomics Can Improve Outcomes in Communication Disorders. Am J Speech Lang Pathol. 2023 Jul 10;32(4):1397-1412. doi: 10.1044/2023_AJSLP-22-00205. Epub 2023 May 5. PMID 37146603
- [Result] Potter NL, VanDam M, Bruce L, Davis J, Eng L, Finestack L, Heinlen V, Scherer N, Schrock C, Seltzer R, Stoel-Gammon C, Thompson L, Peter B. Virtual Post-Intervention Speech and Language Assessment of Toddler and Preschool Participants in Babble Boot Camp. J Speech Lang Hear Res. 2024 Sep 26;67(9S):3327-3339. doi: 10.1044/2023_JSLHR-22-00687. Epub 2023 May 26. PMID 37235746